CLINICAL TRIAL: NCT06933134
Title: Prospective Validation of a Pharmacological Biomarker for Low-Dose Rituximab in Rheumatoid Arthritis
Acronym: PROLOD-RA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230304 - PROLOD-RA
Record Dates: First submitted 2025-03-25; First posted 2025-04-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: pharmacological biomarker; rituximab; retreatment; low dose
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 blood samples at months 0, 3, 6, 9 and 12
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients group: The number of subjects required for our study was set at 30. It's a single-centre prospective non-interventional descriptive study. Patients will be followed every 3 months during 12 months. At inclusion, they will receive a first cycle of low-dose rituximab followed by a second cycle at 6 months.

SUMMARY:
Evaluation of the prediction of clinical response to rituximab at a dose of 1000 mg once using a pharmacological model including several pharmacokinetic and pharmacodynamic parameters.

DETAILED DESCRIPTION:
Rituximab is an anti-CD20 monoclonal antibody which is effective in RA. The dose indicated in the marketing authorisation is 1000 mg twice per cycle. However, rituximab is associated with adverse events, and more specifically the risk of infection, which seems to be dose-dependent. The dose of 1000 mg once a cycle has been evaluated and is non-inferior for maintenance treatment. Lower doses than 1000 mg once could also be sufficient, but there is a lack of predictive criteria to guide clinicians in their search for the minimal effective dose for a given patient.

In our center, a PK-PD model including several parameters (body surface area, serum IgG concentration, residual rituximab concentrations and CD4+ T-cell count) has enabled to quantify part of the concentration-effect relationship of rituximab in this indication and at standard dose (1000 mg twice at 15-day intervals). On the basis of this model, a model for predicting clinical response has been developed.with reliable prediction of clinical response.

The aim of this study is to apply this model to patients receiving low-dose rituximab (1000 mg once per cycle) and to evaluate the prediction of clinical response to low-dose rituximab using this model.

Correlation and coefficient of determination between DAS28-CRP observed 6 months after a second low-dose cycle and DAS-28 predicted by a PK-PD model taking into account gender, body surface area, IgG concentration, rituximab concentration and CD4 T-cell count.

ELIGIBILITY:
Inclusion Criteria:

. Age ≥ 18 years

* Diagnosis of rheumatoid arthritis meeting ACR/EULAR 2010 criteria.
* Candidates for a Low Dose regimen: on standard dose rituximab and with a good clinical response according to the referring rheumatologist. No maximum duration of use of standard-dose rituximab has been defined.
* In the case of co-prescription of csDMARDs (Methotrexate, Leflunomide, Salazopyrine, Plaquenil), the dose must have been stable for 3 months.
* If corticosteroids are co-prescribed, the dose should be ≤ 10 mg/d and stable for 3 months.

Exclusion Criteria:

* Other associated targeted disease-modifying therapy
* Sjögren's syndrome or other associated inflammatory rheumatism
* Fibromyalgia or other pathology having an impact on the assessment of disease activity
* Any active haematological disease affecting lymphocytes (chronic lymphocytic leukaemia, Hodgkin's and non-Hodgkin's lymphomas, lymphoplasmacytic lymphoma, T lymphoma).
* Opposition to data processing
* No inclusion of persons covered by articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code (e.g. minors, protected adults, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of rheumatoid arthritis meeting ACR/EULAR 2010 criteria on standard-dose rituximab with a good clinical response.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Observed Disease Activity Score(DAS) 28-CRP | 6 months after a second low-dose cycle
  DAS28-CRP measured by the clinician 6 months after the second cycle of rituximab
Calculated DAS28-CRP | 6 months after a second low-dose cycle
  DAS28-CRP calculated 6 months after the second cycle of rituximab by a PK-PD model, taking into account gender, body surface area in m2, IgG concentration, rituximab concentration and CD4+ T-cell count

SECONDARY OUTCOMES:
Prevalence observed DAS28-CRP | 3 months and 6 months of the first and second cycle of low-dose rituximab
  * Percentage of patients with a DAS28-CRP < 3.2 at 3 months and 6 months of the first and second cycle of low-dose rituximab
  * Percentage of patients with a DAS28-CRP <2.6 at 3 months and 6 months of the first and second cycle of low-dose rituximab
Description of events | From enrolment to 12 months
  Description of moderate and severe infectious events. Description of adverse events occurring during infusions
prevalence calculated DAS28-CRP | 6 months of the second cycle of low-dose rituximab
  * percentage of patients with a predicted DAS 28 CRP < 3.2 at 6 months of the second cycle of low-dose rituximab
  * percentage of patients with a predicted DAS 28 CRP < 2.6 at 6 months of the second cycle of low-dose rituximab
CD4 T cell count | 6 months of a second cycle of low dose rituximab.
  T cell count (< 500/mm3)
immunoglobulin G level | 6 months of a second cycle of low dose rituximab.
  immunoglobulin G level (< 6 g/L)

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided